CLINICAL TRIAL: NCT02560948
Title: A Multicenter, International, Randomised, Double-blind, Placebo Controlled Study to Demonstrate the Clinical Efficacy and Safety of a Subcutaneous Immunotherapy With gpASIT+™ in Patients With Grass Pollen-induced Allergic Rhinoconjunctivitis
Brief Title: Clinical Efficacy and Safety of a Subcutaneous Immunotherapy With gpASIT+™ in Patients With Grass Pollen-induced Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioTech Tools S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTT-gpASIT009
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2015-09

CONDITIONS: Hay Fever
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo solution
- gpASIT+TM (Experimental)
  Interventions: Biological: gpASIT+TM

INTERVENTIONS:
Biological: Placebo solution — 4 x 2 injections over 21 days
  Arms: Placebo
Biological: gpASIT+TM — 4 x 2 injections over 21 days
  Arms: gpASIT+TM

SUMMARY:
gpASIT+TM product is based on highly purified allergen fragments obtained from grass pollen. The purpose of this study is to demonstrate the clinical efficacy and safety of a subcutaneous immunotherapy with gpASIT+™ in patients with grass pollen-induced allergic rhinoconjunctivitis compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Allergy diagnosis:

  * A medical history of moderate to severe seasonal allergic rhinoconjunctivitis (SARC) for the grass pollen season during at least the two previous seasons (definition of allergy severity according to ARIA (Bousquet et al 2001))
  * A positive skin prick test (SPT - wheal diameter ≥ 3 mm) to grass pollen mixture, histamine wheal ≥ 3 mm, NaCl control reaction < 2 mm
  * Specific IgE against grass pollen (with recombinant allergens - g213) > 0.7 kU/L
  * Positive response to CPT with at least 10,000 SQ-E/mL of grass allergens
* Patients treated with anti-allergic medication for at least 2 grass pollen seasons prior to enrollment
* For asthmatic patients: confirmed diagnosis of controlled asthma according to Global Initiative for Asthma (GINA) guidelines (steps 1-3, GINA 2014)

Key Exclusion Criteria:

* Previous immunotherapy with grass allergens within the last 5 years
* Ongoing immunotherapy with grass allergens or any other allergens
* Patients with a history of anaphylaxis, including food (e.g. peanut or marine animals) or hymenoptera venom (e.g. bee or wasp stings) or medication (e.g. penicillin)
* Patients with partly controlled or uncontrolled asthma according to GINA guidelines (GINA 2014)
* Patients with chronic asthma or emphysema, particularly with a forced expiratory volume in 1 second (FEV1) < 80% of the predicted value (ECSC) or with a peak expiratory flow (PEF) < 70% of the individual optimum value
* Patients symptomatic to inhaled allergens circulating during the grass pollen season (specific to each country: e.g. birch, hazel, mugwort, ragweed, olive, Alternaria alternata)
* Patients symptomatic to perennial inhaled allergens (house dust mites, cat, dog) to which the patients are regularly exposed

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 554 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Combined Symptom and Medication Score (CSMS) | over the peak (corresponding to 14 consecutive days with highest pollen counts) of grass pollen season estimated between 3 and 6 months after treatment

SECONDARY OUTCOMES:
Combined Symptom and Medication Score (CSMS) | over the entire grass pollen season estimated between 3 and 6 months after treatment
Symptom sub-scores (Eyes, Nose) | over the peak period (14 consecutive days with highest pollen counts within grass pollen season) and over the pollen season estimated between 3 and 6 months after treatment
Well days: number of days with symptomatic score below or equal to 2 and no rescue medication | over the peak period (14 consecutive days with highest pollen counts within grass pollen season) and over the pollen season estimated between 3 and 6 months after treatment
Lung Symptom Score (LLS: the average of coughing, wheezing, chest tightness and exercise induced dyspnoea scores) in asthmatic patients | over the peak period (14 consecutive days with highest pollen counts within grass pollen season) and over the pollen season estimated between 3 and 6 months after treatment
Total Symptom Score (TSS: the sum of the nose, eye and lung scores) in asthmatic patients | over the peak period (14 consecutive days with highest pollen counts within grass pollen season) and the pollen season estimated between 3 and 6 months after treatment
Use of rescue medication to relief asthma symptoms in asthmatic patients | over the peak period (14 consecutive days with highest pollen counts within grass pollen season) and the pollen season estimated between 3 and 6 months after treatment
Conjunctival Provocation Test (CPT) outcomes | at baseline and up to 6 weeks
Standardized Quality-of-Life Questionnaires for asthma and rhinoconjunctivitis | between 2 weeks and 8 months after treatment
Number of working day lost due to grass pollen induced-allergy symptoms | between 2 weeks and 8 months after treatment
Loss of productivity at work due to grass pollen induced-allergy symptoms, using a visual analog scale (VAS) | between 2 weeks and 8 months after treatment
Solicited adverse events | up to 4 weeks
  * Local reactions at the injection site (swelling and redness)
  * Allergic systemic reactions
Unsolicited adverse events and serious adverse events | up to 8 months
Physical examinations and vital signs | up to 8 months
Laboratory investigations (haematology, clinical biochemistry, immunological parameters) | up to 8 months
Use of rescue medication | up to 4 weeks

OTHER OUTCOMES:
Production of grass pollen specific immunoglobulins IgE, IgG and IgG4 | up to 8 months
Production of blocking antibodies (FAB assay) | up to 8 months
Reduction of Th2 response by measuring IL-4+ and IFN-gamma+ production | up to 8 months
Induction of regulatory T cells (Treg) | up to 8 months
Induction of regulatory B cells (Breg) and their phenotyping | up to 8 months
Reduction of basophil activation measured through detection of CD63 expression marker on activated cells | up to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mösges, Professor, Principal Investigator — Private practice, Aachen, Germany; Claus Bachert, Professor, Principal Investigator — UZ Gent, Gent, Belgium; Petr Panzner, MD, Principal Investigator — University Hospital of Pilsen, Pilsen, Czech Republic; Frédéric de Blay, Professor, Principal Investigator — CHRU de Strasbourg, Strasbourg, France; Enrico Iemoli, MD, Principal Investigator — Clinica dell'Azienda Ospedaliera Luigi Sacco Di Milano, Milano, Italy; Joachin Sastre, Professor, Principal Investigator — Fundación Jiménez Díaz, Madrid,Spain
Locations (3):
- University Hospital Ghent, Ghent, Belgium
- Clinica dell'Azienda Opsedaliera Luigi Sacco, Milan, Italy
- Fundacion Jiménez Diaz, Madrid, Spain

REFERENCES:
- [Derived] Sharif H, Singh I, Kouser L, Mosges R, Bonny MA, Karamani A, Parkin RV, Bovy N, Kishore U, Robb A, Katotomichelakis M, Holtappels G, Derycke L, Corazza F, von Frenckell R, Wathelet N, Duchateau J, Legon T, Pirotton S, Durham SR, Bachert C, Shamji MH. Immunologic mechanisms of a short-course of Lolium perenne peptide immunotherapy: A randomized, double-blind, placebo-controlled trial. J Allergy Clin Immunol. 2019 Sep;144(3):738-749. doi: 10.1016/j.jaci.2019.02.023. Epub 2019 Mar 5. PMID 30844425